CLINICAL TRIAL: NCT04344002
Title: Observational Retrospective Register of Spanish Lung and Melanoma Cancer Patients With COVID19 Disease
Brief Title: LunG and Melanoma canceR pAtients coVId19 Disease (GRAVID)
Acronym: GRAVID
Status: Completed | Type: Observational
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Other Study IDs: GECP 20/02_GRAVID
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Covid-19; Lung Cancer
Keywords: covid-19; coronavirus; lung cancer
MeSH Terms: conditions — COVID-19; Lung Neoplasms; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lung cancer+COVID-19: lung cancer patients diagnosed with COVID-19

SUMMARY:
This is a multi-centre study on lung cancer patients which experienced COVID-19. Information on clinical features, clinical course, management and outcomes will be collected for both, thoracic cancers and COVID-19 infection. Firstly, investigators will be registered in an online secure registry. After that, a protocol will be developed in order to collect clinical data for the research. It will also include I on the care organization or the perception of the patient and their family members.

The final stage will consist on retrospective data collection from patients. So, it is a retrospective study data collection, preceded by prospective data registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with lung cancer
* Patients who have contracted COVID-19 infection

Exclusion Criteria:

* Patients diagnosed with lung cancer but no confirmation of COVID-19 infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with lung cancer and who have been infected with COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 886 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Clinical data of lung cancer patients with COVID-19 diagnoses | From the diagnosis of the COVID until the patient is cured or dies, whichever comes first, assessed up to 5 years
  Describe characteristics and evolution of Spanish patients preferably with lung cancer who contract COVID 19 infection with identification and study of factors of interest, as well as clinical data.
Diagnosis data | From the diagnosis of the COVID until the patient is cured or dies, whichever comes first, assessed up to 5 years
  Describe characteristics and evolution of Spanish patients preferably with lung cancer who contract COVID 19 infection with identification and study of factors of interest, as well as data about diagnosis
Treatments received | From the diagnosis of the COVID until the patient is cured or dies, whichever comes first, assessed up to 5 years
  Describe characteristics and evolution of Spanish patients preferably with lung cancer who contract COVID 19 infection with identification and study of factors of interest, as well as treatments received
Prognostic factors | From the diagnosis of the COVID until the patient is cured or dies, whichever comes first, assessed up to 5 years
  Describe characteristics and evolution of Spanish patients preferably with lung cancer who contract COVID 19 infection with identification and study of factors of interest, as well as prognostic factors.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano MD Provencio, MD, Study Chair — Hospital Puerta de Hierro de Majadahonda de Madrid; Cristina MD Avendaño Solá, MD, Study Chair — Hospital Puerta de Hierro de Majadahonda de Madrid; María MD González-Cao, MD, Study Chair — Hospital Universitario Dexeus de Barcelona.
Locations (75):
- Spain (75):
  - Complejo Hospitalario Universitario de Ferrol, Ferrol, A Coruña
  - H. Clínica Benidorm, Benidorm, Alicante
  - Hospital de Elche, Elche, Alicante
  - Hospital General Universitario de Elda, Elda, Alicante
  - Hospital de Torrevieja, Torrevieja, Alicante
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Cetir Centre Mèdic, Esplugues de Llobregat, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Hospital Instituto Onkologikoa, Donostia / San Sebastian, Basque Country
  - Hospital Universitario de Galdakao, Galdakao, Bizkaia
  - Complejo Hospitalario de la Coruña, A Coruña, Coruña
  - H. Insular de Gran Canarias, Las Palmas de Gran Canaria, Gran Canarias
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Severo Ochoa, Leganés, Madrid
  - Hospital Universitario de Móstoles, Móstoles, Madrid
  - Hospital de Manacor, Manacor, Mallorca
  - Hospital Costa del Sol, Marbella, Málaga
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Sant Joan de Reus, Reus, Tarragona
  - Hospital Verge de la Cinta, Tortosa, Tarragona
  - H. Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Universitario de La Ribera, Alzira, Valencia
  - Hospital de Manises, Manises, Valencia
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital de Basurto, Bilbao, Vizcaya
  - H. Gen. Universitario Alicante, Alicante
  - Hospital Ntra. Sra. Sónsoles, Ávila
  - H. Universitario Quirón Dexeus, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - H. Duran i Reynals-ICO, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario de Puerto Real, Cadiz
  - Hospital La Mancha Centro, Ciudad Real
  - Hospital Virgen de la Luz, Cuenca
  - Hospital Dr. Josep Trueta, Girona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital de Guadalajara, Guadalajara
  - Complejo Asistencial Universitario de León, León
  - Hospital San Millan Y San Pedro, Logroño
  - Hospital Universitario Lucus Augusti, Lugo
  - MD Anderson, Madrid
  - H.U. Puerta de Hierro, Madrid
  - Fundación Jimenez Diaz, Madrid
  - Hospital Universitario Infanta Sofía, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital de Sanchinarro, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Universitario del Henares, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Santa María Naí, Ourense
  - Hospital Son Espases, Palma de Mallorca
  - H. Son Llàtzer, Palma de Mallorca
  - Hospital Clinico de Salamanca, Salamanca
  - Hospital universitario Nuestra Señora Candelaria, Santa Cruz de Tenerife
  - Hospital General de Segovia, Segovia
  - Hospital Virgen del Rocío, Seville
  - Hospital Sant Pau i Santa Tecla, Tarragona
  - H. General U. de Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Dr. Peset, Valencia
  - Hospital Politècnic i Universitari La Fe, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - H. Miguel Servet, Zaragoza
  - Hospital Universitario de Áraba, Vitoria-Gasteiz, Áraba

REFERENCES:
- [Derived] Gonzalez-Cao M, Puertolas T, Martinez-Vila C, Carrera C, Maldonado Seral C, Rodriguez-Jimenez P, Sequero S, Cerezuela-Fuentes P, Feltes Ochoa R, Munoz E, Antonanzas Basa M, Martin-Liberal J, Soria A, Francisco Rodriguez Moreno J, Marquez-Rodas I, Lopez Criado P, Luis Manzano J, Lopez-Castro R, Ayala de Miguel P, Villalobos L, Martin Algarra S, Gonzalez-Barrallo I, Boada A, Garcia Castano A, Puig S, Crespo G, Luna Fra P, Aguayo Zamora C, Feito Rodriguez M, Valles L, Drozdowskyj A, Gardeazabal J, Antonio Fernandez-Morales L, Rodrigo A, Cruz R, Yelamos O, Rubio B, Mujica K, Provencio M, Berrocal A; Spanish Melanoma Group (GEM). SARS-CoV-2 infection in patients with melanoma: results of the Spanish Melanoma Group registry. Clin Transl Oncol. 2023 Mar;25(3):768-775. doi: 10.1007/s12094-022-02985-7. Epub 2022 Dec 24. PMID 36566266
- See also: Web page of the sponsor where users can find more information about Fundacion GECP studies — http://www.gecp.org